CLINICAL TRIAL: NCT02066519
Title: Benefits and Tolerance of Exercise in Patients With Generalized and Stabilized Myasthenia Gravis
Acronym: MGEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P111106
Record Dates: First submitted 2014-01-13; First posted 2014-02-19 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia gravis; physical exercise; quality of life; muscular performance; fatigability
MeSH Terms: conditions — Myasthenia Gravis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise arm (Experimental): Arm with physical exercise on rowing machine between M3 and M6
  Interventions: Behavioral: Physical exercise programme using a rowing machine
- Control arm (No Intervention): Arm with standard medical care without additional physical exercise

INTERVENTIONS:
Behavioral: Physical exercise programme using a rowing machine — 3 sessions per week of individualized physical training using a rowing machine during 3 months.
  Arms: Physical exercise arm

SUMMARY:
The purpose of this study is to demonstrate that a 3 months physical exercise programme improves the Quality of Life of patients with generalized Myasthenia Gravis (MG) stabilized since at least 6 months under prednisone and/or azathioprine.

DETAILED DESCRIPTION:
Three centers randomized simple blind clinical trial whose objective is to assess the efficacy on QoL improvement, and the tolerance of physical exercise over a period of 3 months in patients with generalized MG who have been stabilized since at least 6 months.

During the 3 months pre-inclusion phase, the characteristics of MG will be collected. Physical activity and performance will be assessed monthly.

MGQOL15 will be assessed at inclusion.

Patients will be randomized in either intervention arm or control arm.

The intervention arm will consist of three sessions exercise per week during three months. The daily exercise will be performed on a rowing machine that will be adapted to the patient's own physical ability.

Physical activity will be measured with the help of an actimeter.

Once a month, MG evolution and tolerance to exercise will be assessed and MG treatment dose will be collected.

Exercise will be interrupted in case of MG exacerbation.

Quality of life and psychological status will be assessed at 3, 6 and 9 months.

Plasma levels of pro and anti-inflammatory cytokines will be measured at 3, 6 and 9 months in order to assess the effects of exercise on immune response.

Patients enrolled in the control arm will benefit from the same follow-up but will not have exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with generalized MG of stage II or III according to the MGFA classification, stabilized for at least 6 months. Criteria for MG are either

   * positive dosage of ant-RACh or MuSK auto-antibodies;
   * If absent, myasthenic symptoms decrement> 10% in EMNG and test the positive prostigmine
2. Patient ≥ 18 and ≤ 70 years old
3. Patient having an health insurance
4. Informed written consent

Exclusion Criteria:

1. Patients under particular protection
2. Enrolment in another biomedical research in the last 3 months;
3. Patients for whom physical practice is contra-indicated because of :

   * Unstable coronary Syndrome or myocardial infarction within the past 3 months
   * Heart failure with systolic ejection fraction < 50 %
   * Respiratory failure defined by a vital capacity (CV) < 70 %
   * Stroke
   * Other neuromuscular pathology
   * Disabling Rheumatologic disease (> 80 % disability according to the Barthel scale)
   * Chronic Pain or disabling orthopaedic conditions
   * Hospitalization in the last 3 months for a serious medical or surgical condition
   * Anemia (hematocrit < 30%)
4. MGFA grade I, grade IV or V
5. Severe cognitive impairment
6. MGQOL-15 below 15/60

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Change in the quality of life between M3 and M6 by MGQOL score | M3 and M6

SECONDARY OUTCOMES:
Muscular strength | M3, M6 and M9
  Muscular strength (before exercise period, after exercise period and 3 months after)
Frequency of MG exacerbations | 6 MONTHS
Frequency and severity of cardiovascular side-effects | 6 MONTHS
Cumulative dose of steroids within the 3 months of the exercise programme | 6 MONTHS
Doses of anticholinesterasic and steroids at 3, 6 and 9 months | M3, M6 and M9
Psychological status (STAI, BECK, MINI et SEI scales) at 3, 6 and 9 months | M3, M6 and M9
Plasma levels of pro- and anti-inflammatory cytokines at 9 months | M9
Muscular fatigability | M3, M6 and M9
  fatigability (before exercise period, after exercise period and 3 months after)
Muscular endurance | M3, M6 and M9
  muscular endurance (before exercise period, after exercise period and 3 months after)
Severity of MG exacerbations | 6 MONTHS
Frequency and severity of respiratory side-effects | 6 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Tarek SHARSHAR, MD, PhD, Principal Investigator — ICU and medical surgery Service, Raymond Poincaré Hospital, 92380 Garches, France
Locations (1):
- ICU and medical surgery department, Raymond Poincaré Hospital, Garches, Hauts-de-Seine, France

REFERENCES:
- [Derived] Birnbaum S, Porcher R, Portero P, Clair B, Demeret S, Eymard B, Gargiulo M, Louet E, Berrih-Aknin S, Le Panse R, Aegerter P, Hogrel JY, Sharshar T; MGEX Study Group. Home-based exercise in autoimmune myasthenia gravis: A randomized controlled trial. Neuromuscul Disord. 2021 Aug;31(8):726-735. doi: 10.1016/j.nmd.2021.05.002. Epub 2021 May 27. PMID 34304969
- [Derived] Birnbaum S, Hogrel JY, Porcher R, Portero P, Clair B, Eymard B, Demeret S, Bassez G, Gargiulo M, Louet E, Berrih-Aknin S, Jobic A, Aegerter P, Thoumie P, Sharshar T; MGEX Study Group. The benefits and tolerance of exercise in myasthenia gravis (MGEX): study protocol for a randomised controlled trial. Trials. 2018 Jan 18;19(1):49. doi: 10.1186/s13063-017-2433-2. PMID 29347991